CLINICAL TRIAL: NCT02634255
Title: The Prospective Randomized Comparison of the Onset Time of Rocuronium in Patients Undergoing Emergency and Elective Surgery
Brief Title: The Onset Time of Rocuronium in Emergency and Elective Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gamze GULGUN, Md, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rocuronium onset
Record Dates: First submitted 2015-12-12; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Inguinal Hernia; Acute Appendicitis
Keywords: rocuronium; onset time; anxiety
MeSH Terms: conditions — Hernia, Inguinal; Appendicitis; Anxiety Disorders | interventions — Rocuronium; Propofol; Fentanyl; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rocuronium elective surgery (Active Comparator): patients undergoing inguinal herniorrhaphy
  Interventions: Drug: Rocuronium elective surgery; Drug: Propofol; Drug: Fentanyl; Other: Ringer Lactate; Device: Acceleromyography device
- Rocuronium emergency surgery (Experimental): patients undergoing appendectomy
  Interventions: Drug: Rocuronium emergency surgery; Drug: Propofol; Drug: Fentanyl; Other: Ringer Lactate; Device: Acceleromyography device

INTERVENTIONS:
Drug: Rocuronium elective surgery — Rocuronium onset time in patients undergoing inguinal herniorrhaphy
  Other Names: esmeron
  Arms: Rocuronium elective surgery
Drug: Rocuronium emergency surgery — Rocuronium onset time in patients undergoing appendectomy
  Other Names: esmeron
  Arms: Rocuronium emergency surgery
Drug: Propofol
Drug: Fentanyl
Other: Ringer Lactate
Device: Acceleromyography device
  Other Names: TOF Guard Sx

SUMMARY:
Rocuronium, a nondepolarizing neuromuscular blocking agent, is used in general anesthesia to provide conditions for endotracheal intubating. Recommended dose is 0,6 mg/kg and 90 seconds after intravenous injection, patients can be intubated.

Anxiety levels may vary in patients undergoing emergency and elective surgery. Patients undergoing emergency surgery may display exaggerated laryngoscopic responses. The purpose of this study is to investigate the effect of patient anxiety levels on the onset time of rocuronium in terms of anxiety scores and train of four (TOF) 0.1 times.

DETAILED DESCRIPTION:
After obtaining ethics committee approval, American Society of Anesthesiologists physiological status 1 (ASA 1) patients, undergoing elective inguinal hernia repair and acute appendectomy, will be included to trial.

Patients will be taken to the operating room without premedication. Spielberger's State-Trait Anxiety Inventory (STAI) will be administered to patients for determining anxiety level.

Electrocardiogram, blood pressure and peripheric oxygen saturation (SpO2) will be monitored. After opening intravenous access on hand dorsum, ringer lactate solution will be given. Neuromuscular monitoring and drug injections will be done as described in "Good Clinical Research Practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents".

TOF-Guard SX acceleromyograph (Organon-Teknika) will be monitored on corrugator supercilii muscle because of its sensitivity to laryngeal muscles. In induction of anesthesia, propofol 2 mg kg-1 and fentanyl 1 mcg kg-1 will be administered intravenously. After loss of conscious, TOF-Guard SX will be calibrated and then 0.6 mg kg-1 rocuronium will be administered in 5 seconds. 20 milliampere (mA) current TOF stimulation (200 ms, square wave, 2 Hz for 1.5 s) will be repeated in every 15 s. Patients will be intubated in TOF 0.1 time.

STAI score, heart rate, systolic blood pressure, diastolic blood pressure, mean arterial pressure, SpO2, TOF 0.1 time and intubation conditions will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18,5-24,9
* ASA 1

Exclusion Criteria:

* Allergy to used drugs during anesthesia
* Neuromuscular disease
* Liver and kidney failure
* Heart failure
* Anticipated difficult airway
* Using aminoglycosides
* BMI<18,5 and BMI>25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Train of Four Ratio (TOF 0.1) | 90 seconds after induction
anxiety score | 15 minutes before induction

CONTACTS AND LOCATIONS:
Overall Officials: Murat Sayın, Assoc Prof, Study Chair — Diskapi Yildirim Beyazit Education and Research Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Plaud B, Debaene B, Donati F. The corrugator supercilii, not the orbicularis oculi, reflects rocuronium neuromuscular blockade at the laryngeal adductor muscles. Anesthesiology. 2001 Jul;95(1):96-101. doi: 10.1097/00000542-200107000-00019. PMID 11465590